CLINICAL TRIAL: NCT06854029
Title: Optimizing Long-Acting Pre-Exposure Prophylaxis and Medications for Opioid Use Disorder Interventions in Carceral Settings
Brief Title: NOTRE: Optimizing Long-Acting Pre-Exposure Prophylaxis and Medications for Opioid Use Disorder Interventions in Carceral Settings
Acronym: NOTRE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Friends Research Institute, Inc. (Other); The Miriam Hospital (Other); University of Arkansas (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00117590; R61DA060583 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections; Opioid Use Disorder; Incarceration; Lens
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders | interventions — cabotegravir; Buprenorphine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups; 1) Daily oral medications for HIV prevention and MOUD treatment, and 2) Long-acting injectable HIV prevention and MOUD treatment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily Oral Pill Arm (Active Comparator): Participants assigned to this arm will be administered daily oral pre-exposure prophylaxis for HIV prevention, as well as daily oral buprenorphine for opioid use disorder
  Interventions: Drug: Cabotegravir Pill; Drug: Buprenorphine Pill
- Long Acting Injectable Arm (Experimental): Participants assigned to this arm will be administered the-long acting injectable formulation of pre-exposure prophylaxis every 1-2 months, as well as the long-acting injectable formulation of buprenorphine, at the same clinic visit.
  Interventions: Drug: Cabotegravir Injection; Drug: Buprenorphine injection

INTERVENTIONS:
Drug: Cabotegravir Injection — Long-acting injection (LAI) Prep + X-RB treatment initiated in jail or prison.
  Arms: Long Acting Injectable Arm
Drug: Cabotegravir Pill — Oral PrEP + SL-B treatment initiated in jail or prison.
  Arms: Daily Oral Pill Arm
Drug: Buprenorphine injection — Long-acting injection (LAI) Prep + X-RB treatment initiated in jail or prison.
  Arms: Long Acting Injectable Arm
Drug: Buprenorphine Pill — Oral PrEP + SL-B treatment initiated in jail or prison.
  Arms: Daily Oral Pill Arm

SUMMARY:
The investigators plan to conduct an R61/33 hybrid type 2 implementation-effectiveness trial that includes 1) a one-year exploratory R61 phase that will enable the development of the intervention protocol needed for the R33 trial phase including concrete R61 phase milestones; 2) a four-year R33 phase that will include a concurrent implementation evaluation and a randomized control trial.

DETAILED DESCRIPTION:
Study aims are: Aim 1 (R61): Develop the intervention protocol for delivery of LAI PrEP + XR-B. We will conduct interviews with stakeholders (staff at partner and other carceral and community sites, n=18:) and currently or recently incarcerated individuals (n=18). Interviews will focus on how to optimize intervention components for the R33 phase. Aim 2 (R33): Evaluate implementation facilitation as a strategy to support co-located LAI PrEP + XR-B in carceral and re-entry settings. Guided by the Consolidated Framework for Implementation Research (CFIR), implementation outcomes from Proctor et al.,including acceptability, appropriateness, adoption, feasibility, and sustainability will be assessed using surveys, interviews, and administrative records. Aim 3 (R33): Compare the effectiveness of co-located LAI PrEP + XR-B to oral PrEP + SL-B. An open-label design will randomly assign 300 adults who are clinically indicated for both PrEP and MOUD and soon-to-be-released from a carceral setting to either LAI Prep + X-RB (n=150) or oral PrEP + SL-B (n=150) treatment initiated in jail or prison. A baseline assessment will be conducted prior to release followed by monthly follow-up for 7 months and a final long-term follow-up visit at 12-months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18) at a participating carceral site;
2. Eligible for release within 120 days (sentenced and/or pretrial). Individuals who might be sentenced to federal prison will be excluded;
3. History of OUD (meeting DSM-5 criteria of moderate or severe opioid use disorder at the time of incarceration; individuals not meeting the opioid-disorder criterion will be eligible if they were treated in an opioid agonist treatment program during the year before incarceration or met OUD criteria in the year prior to incarceration);
4. HIV negative (as confirmed by a HIV rapid test);
5. Clinically indicated for PrEP based on CDC guidelines during incarceration and/or the year prior to incarceration;
6. Willing to enroll in buprenorphine treatment and PrEP and be randomized to either study arm; and
7. Report that, during community re-entry they will reside in the geographic locations of the study.

Exclusion Criteria:

1. Liver function test levels greater than four times normal (if we are unable to obtain labs, a determination by our site partner physicians will be made to allow inclusion);
2. Active medical illness that may make participation hazardous (e.g., unstable diabetes, heart disease; renal impairment, Hepatitis B);
3. Conditions or medications that may predispose to QTc prolongation (personal or family history of long QT syndrome, hypokalemia, medications that prolong QTc interval, e.g., macrolide antibiotics, azole antifungal compounds, anti-arrhythmics, antipsychotics and antidepressants);
4. Untreated psychiatric disorder that may make participation hazardous (e.g., untreated psychosis, treated psychiatric disorders will be allowed);
5. Known allergic reaction to PrEP or buprenorphine; and
6. Suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
PrEP adherence, time to dropout | up to 12 months
  Dropout is defined as missing treatment for 7 consecutive days.
Buprenorphine adherence, time to dropout | up to 12 months
  Dropout is defined as missing treatment for 7 consecutive days.

SECONDARY OUTCOMES:
Substance use as measured by number of participants with positive Urine Drug Test (UDT) | up to 12 months
Number of participants with a fatal or non-fatal overdose | up to 12 months
Number of participants engaging in HIV risk behaviors | up to 12 months
Number of participants with past criminal system engagement | Baseline
Number of participants with HIV acquisition | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Brinkley-Rubinstein, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Our data and research findings will be shared with other researchers through the customary means of peer-reviewed publications and at national and international conferences and symposia, such as the annual meeting of the Academic Consortium on Criminal Justice Health, the American Public Health Association.
  We will ensure that publications reporting on study data and results will be made available to interested scientists by submitting an electronic version of all papers, upon acceptance for publication, to the National Library of Medicine's PubMed Central.
  In addition, we will cite this grant in any products emanating from this research study. Whenever possible, we will make resulting publications open access. In addition, our team, whenever possible, will make the data underlying the conclusions of peer-reviewed scientific research publications freely available in public repositories at the time of initial publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Scientific data will be made available after all longitudinal data is collected (baseline, follow-up data) and has undergone rigorous quality control. In addition, data will be made available after the primary outcome papers are accepted for publication. An exception to this will be sharing more routinely with the HIV/Justice Research Network Data Coordination Center.